CLINICAL TRIAL: NCT05478720
Title: DON in Pediatric Cerebral Malaria: A Phase I/IIa Dose-Escalation Safety Study
Brief Title: DON in Pediatric Cerebral Malaria
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Douglas Postels, MD, MS (Unknown)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Douglas Postels, Professor of Pediatric Neurology, Children's National Research Institute
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21/04/2676; 21-0005 (Other: DMID); PAR-18-633 (Other Grant/Funding Number: DMID)
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Malaria, Cerebral
Keywords: malaria; Plasmodium falciparum
MeSH Terms: conditions — Malaria, Cerebral; Malaria; Malaria, Falciparum | interventions — Diazooxonorleucine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Part 1: Adult groups Healthy / Uncomplicated Malaria - Groups of 10 adult participants will be enrolled sequentially, with safety assessment and dose escalation for each group if safety criteria are satisfied in the previous group.
  Pediatric Arm: Enrollment of pediatric participants will begin if safety criteria are satisfied in adults previously enrolled. The pediatric study will be randomized and placebo-controlled with DON or Placebo doses added to standard of care therapy. Interim assessments are planned to determine dosing for subsequent participants.
Masking Description: Part 1: None (Open Label) Part 2: Blinded (Participants/ Caregivers, Study Staff)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (13):
- Dose escalation in healthy Malawian adults - 0.1 mg/kg IV DON (Experimental): The first 10 healthy adult participants enrolled will receive a single 0.1 mg/kg intravenous (IV) DON. If this dose is proven safe, in each subsequent group of 10, the dose will be increased to 1.0 mg/kg IV DON and then 5.0 mg/kg IV DON the final group will receive 10.0 mg/kg IV DON.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in healthy Malawian adults - 1.0 mg/kg IV DON (Experimental): The first 10 healthy adult participants enrolled will receive a single 0.1 mg/kg intravenous (IV) DON. If this dose is proven safe, in each subsequent group of 10, the dose will be increased to 1.0 mg/kg IV DON and then 5.0 mg/kg IV DON the final group will receive 10.0 mg/kg IV DON.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in healthy Malawian adults - 5.0 mg/kg IV DON (Experimental): The first 10 healthy adult participants enrolled will receive a single 0.1 mg/kg intravenous (IV) DON. If this dose is proven safe, in each subsequent group of 10, the dose will be increased to 1.0 mg/kg IV DON and then 5.0 mg/kg IV DON the final group will receive 10.0 mg/kg IV DON.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in healthy Malawian adults - 10.0 mg/kg IV DON (Experimental): The first 10 healthy adult participants enrolled will receive a single 0.1 mg/kg intravenous (IV) DON. If this dose is proven safe, in each subsequent group of 10, the dose will be increased to 1.0 mg/kg IV DON and then 5.0 mg/kg IV DON the final group will receive 10.0 mg/kg IV DON.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in Malawian adults with uncomplicated malaria - 0.1 mg/kg IV DON (Experimental): The first 10 adults with uncomplicated malaria participants enrolled will receive a single 0.1 mg/kg intravenous (IV) DON. If this dose is proven safe, in each subsequent group of 10, the dose will be increased to 1.0 mg/kg IV DON and then 5.0 mg/kg IV DON, and then the final group will receive 10.0 mg/kg IV DON.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in Malawian adults with uncomplicated malaria - 1.0 mg/kg IV DON (Experimental): The first 10 adults with uncomplicated malaria participants enrolled will receive a single 0.1 mg/kg intravenous (IV) DON. If this dose is proven safe, in each subsequent group of 10, the dose will be increased to 1.0 mg/kg IV DON and then 5.0 mg/kg IV DON, and then the final group will receive 10.0 mg/kg IV DON.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in Malawian adults with uncomplicated malaria - 5.0 mg/kg IV DON (Experimental): The first 10 adults with uncomplicated malaria participants enrolled will receive a single 0.1 mg/kg intravenous (IV) DON. If this dose is proven safe, in each subsequent group of 10, the dose will be increased to 1.0 mg/kg IV DON and then 5.0 mg/kg IV DON, and then the final group will receive 10.0 mg/kg IV DON.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in Malawian adults with uncomplicated malaria - 10.0 mg/kg IV DON (Experimental): The first 10 adults with uncomplicated malaria participants enrolled will receive a single 0.1 mg/kg intravenous (IV) DON. If this dose is proven safe, in each subsequent group of 10, the dose will be increased to 1.0 mg/kg IV DON and then 5.0 mg/kg IV DON, and then the final group will receive 10.0 mg/kg IV DON.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in Malawian children with cerebral malaria - 0.1 mg/kg IV DON - Cohort 1 (Experimental): After adult doses are shown to be safe. Of the first 6 children with cerebral malaria enrolled, 4 will receive 0.1 mg/kg IV DON, and 2 will receive placebo.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in Malawian children with cerebral malaria - 0.1 mg/kg IV DON - Cohort 2 (Experimental): 10 participants will receive 0.1 mg/kg IV DON, and 2 will receive placebo.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in Malawian children with cerebral malaria - 1.0 mg/kg IV DON - Cohort 3 (Experimental): 14 participants will receive 1.0 mg/kg IV DON, and 4 will receive placebo.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in Malawian children with cerebral malaria - 0.1 or 1.0 mg/kg IV DON - Cohort 4 (Experimental): 36 participants will receive 0.1 mg/kg IV DON (n=12) or 1.0 mg/kg IV DON (n=12), and 12 will receive placebo.
  Interventions: Drug: 6-diazo-5-oxo-L-norleucine (DON)
- Dose escalation in Malawian children with cerebral malaria - placebo (Placebo Comparator): Cohort 1 will dose 2 participants to receive placebo Cohort 2 will dose 2 participants to receive placebo Cohort 3 will dose 4 participants to receive placebo Cohort 4 will dose 12 participants to receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 6-diazo-5-oxo-L-norleucine (DON) — Single intravenous dose ranging from 0.1-10 mg/kg per dose
  Other Names: NSC 7365
  Arms: Dose escalation in Malawian adults with uncomplicated malaria - 0.1 mg/kg IV DON; Dose escalation in Malawian adults with uncomplicated malaria - 1.0 mg/kg IV DON; Dose escalation in Malawian adults with uncomplicated malaria - 10.0 mg/kg IV DON; Dose escalation in Malawian adults with uncomplicated malaria - 5.0 mg/kg IV DON; Dose escalation in healthy Malawian adults - 0.1 mg/kg IV DON; Dose escalation in healthy Malawian adults - 1.0 mg/kg IV DON; Dose escalation in healthy Malawian adults - 10.0 mg/kg IV DON; Dose escalation in healthy Malawian adults - 5.0 mg/kg IV DON
Drug: Placebo — Single intravenous dose of saline
  Other Names: Saline
  Arms: Dose escalation in Malawian children with cerebral malaria - placebo
Drug: 6-diazo-5-oxo-L-norleucine (DON) — Single intravenous dose ranging from 0.1-1.0 mg/kg per dose
  Other Names: NSC 7365
  Arms: Dose escalation in Malawian children with cerebral malaria - 0.1 mg/kg IV DON - Cohort 1; Dose escalation in Malawian children with cerebral malaria - 0.1 mg/kg IV DON - Cohort 2; Dose escalation in Malawian children with cerebral malaria - 0.1 or 1.0 mg/kg IV DON - Cohort 4; Dose escalation in Malawian children with cerebral malaria - 1.0 mg/kg IV DON - Cohort 3

SUMMARY:
The goal of this clinical trial is to evaluate the safety of a single intravenous dose of DON in healthy adults, adults with uncomplicated malaria, and children 12 months-14 years old with clinically defined Cerebral Malaria. The main objectives are:

* Determine the pharmacokinetic (PK) profile of a single dose of DON in children with CM
* Determine if administration of a single intravenous dose of DON as an adjunctive therapy in children with CM is associated with improved intracerebral blood flow dynamics on transcranial doppler (TCD)
* Determine if administration of a single intravenous dose of DON as an adjunctive therapy in children with CM is associated with a reduction in brain volume score on magnetic resonance imaging (MRI)
* Determine if administration of a single intravenous dose of DON as an adjunctive therapy in children with cerebral malaria is associated with changes in electroencephalogram (EEG) pattern
* Exploratory: Explore the metabolic mechanisms of action of adjunctive DON in children with CM

Healthy adult participants will receive:

* anti-emetic ondansetron
* one dose of DON

Adults with uncomplicated malaria will receive:

* anti-emetic ondansetron
* one dose of DON
* artemisinin-combination therapies per Malawi Ministry of Health guidelines

Pediatric participants will receive:

* one dose of DON
* anti-emetic ondansetron and per Malawi Ministry of Health guidelines:
* enteral lumefantrine-artemether therapy, and
* artesunate therapy

DETAILED DESCRIPTION:
The initial study to be conducted under this IND is a 2 part dose escalation study. The first part contains 2 groups that will be open-label, dose escalation, and will define the safety of 6-diazo-5-oxo-L-norleucine (DON) in African adults (>18 years old), who are healthy or who have uncomplicated malaria.

Each of the two adult groups will enroll 40 participants broken down into 4 dosage groups with safety evaluations before each dose increase. The first 10 participants enrolled will receive 0.1 mg/kg intravenous (IV) DON. If this dose is proven safe, the dose will be increased to 1.0 mg/kg IV DON, and then 5.0 mg/kg IV DON, and then the final group will receive 10.0 mg/kg IV DON. Each adult dosage group contains 10 healthy participants and 10 participants with uncomplicated malaria. The total number of adult participants enrolled is 80 (20 participants at 4 doses). All participants will receive only one dose of DON.

Adult participants will receive a premedication dose of the antiemetic ondansetron, 5 mg IV, administered 30 minutes prior to DON, and repeated 8 and 16 hours later. The duration of study participation for all adult participants is six months.

Part 2 of the study will be a randomized, placebo-controlled, dose-escalation study in children ages 12 months to 14 years with cerebral malaria to determine safety. Pediatric enrollments will span three malaria seasons, which will be carried out in Study Years 3-5, with a planned interim analysis after cohort 3. In cohort 1 we will first enroll 6 sentinel pediatric participants who will receive intravenous artesunate therapy, enteral lumefantrine-artemether therapy, and either adjunctive DON 0.1 mg/kg or placebo randomized 2:1. Cohort 2 will enroll 12 participants who will receive intravenous artesunate therapy, enteral lumefantrine-artemether therapy, and either adjunctive DON 0.1 mg/kg or placebo randomized 5:1.Cohort 3 will enroll 18 participants who will receive intravenous artesunate therapy, enteral lumefantrine-artemether therapy, and either adjunctive DON 1.0 mg/kg or placebo randomized 7:1. Cohort 4 will enroll 36 participants who will receive intravenous artesunate therapy, enteral lumefantrine-artemether therapy, and either adjunctive DON 0.1 mg/kg, DON 1.0 mg/kg or placebo randomized 1:1:1. Pediatric participation in the study will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

For Healthy Adults (Arm 1):

* 18 years and older
* Informed consent obtained and ICF signed
* Temperature ≤ 37.5 °C
* BMI 18.5-25 kg/m2
* Creatinine ≤ 110 mmol/L (≤ 1.2 mg/dL; males) or ≤ 90 mmol/L (≤ 1.0 mg/dL; females)
* Hemoglobin ≥ 7 g/dL or hematocrit/ packed-cell volume (PCV) ≥ 20%
* Thick or thin blood smear negative for asexual forms of P. falciparum
* Negative pregnancy test for persons of child-bearing potential

For Adults with Uncomplicated Malaria (Arm 2):

* 18 years and older
* Informed consent obtained and ICF signed
* Temperature ≥ 38 °C or history of fever in the past 24 hours
* Thick or thin blood smear positive for asexual forms of P. falciparum (parasite count and speciation documented)
* Hemoglobin ≥ 7 g/dL or hematocrit/ PCV ≥ 20%
* BMI 18.5-25 kg/m2
* Creatinine ≤ 110 mmol/L (≤ 1.2 mg/dL; males) or ≤ 90 mmol/L (≤ 1.0 mg/dL; females)
* Glasgow coma score of 15
* Respiratory rate ≤ 20 breaths/ minute
* Oxygen saturation ≥ 90% on room air
* Negative pregnancy test for person of child-bearing potential

For Children with Cerebral Malaria (Arm 3):

* Age 12 months-14 years old
* Informed consent obtained and ICF signed by parent or guardian
* Temperature ≥ 38 °C or history of fever in the last 24 hours
* Thick or thin blood smear positive for asexual forms of P. falciparum
* Blantyre coma score ≤ 2
* No other explanation for coma by history or physical exam
* Hematocrit or PCV ≥ 18%
* Negative pregnancy test for persons of child-bearing potential
* Creatinine ≤ 1.5 mg/dL
* Aspartate aminotransferase (AST) < 280 IU/L
* Alanine aminotransferase (ALT) < 195 IU/L

Exclusion Criteria (All Participants):

* Pregnancy or lactation (participants of child-bearing potential ages 9-59 years will undergo pregnancy testing prior to administration of the intervention)
* Participants attempting to become pregnant
* Currently taking highly active antiretroviral therapy (HAART)
* Currently taking anti-tuberculosis medications
* Allergy to ondansetron

Additional Exclusion Criteria for Children with Cerebral Malaria (Arm 3):

* Cloudy cerebrospinal fluid (indicative of a probable bacterial central nervous system infection)
* Malnutrition defined as a more than or equal to two standard deviations below the mean weight for height and/ or MUAC ≤ 12.5 cm (due to inability to adequately care for children with severe malnutrition on the PRW)
* Allergy to ondansetron or ceftriaxone
* Coma for > 72 hours
* Have taken a CYP3A4 inhibitor within 7 days of enrollment

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of local AEs occurring within 14 days after the administration of DON | 14 days
  Number of AEs
Incidence of systemic AEs occurring within 14 days after the administration of DON | 14 days
  Number of AEs
Incidence of systemic SAEs occurring within 14 days after the administration of DON | 14 days
  Number of SAEs - pediatric arms only

SECONDARY OUTCOMES:
PK measurement of DON in sera of recipients measured by half life | Measured through 18 hours post infusion
  Measurement of half life
PK measurement of DON in sera of recipients measured by volume of distribution | Measured through 18 hours post infusion
  Measurement of Vd
PK measurement of DON in sera of recipients measure by maximum concentration (Cmax) | Measured through 18 hours post infusion
  Measurement of Cmax
PK measurement of DON in sera of recipients measure by time of maximal concentration (Tmax) | Measured through 18 hours post infusion
  Measurement of Tmax
PK measurement of DON in sera of recipients measure by area under the concentrations vs. time curve (AUC) | Measured through 18 hours post infusion
  Measurement of AUC
PK measurement of DON in sera of recipients measure by clearance | Measured through 18 hours post infusion
  Clearance measured over time
PK measurement of DON in sera of recipients measure by elimination rate | Measured through 18 hours post infusion
  Elimination over time
PK measurement of DON in sera of recipients measure by terminal T1/2 | Measured through 18 hours post infusion
  Measurement of terminal T1/2

OTHER OUTCOMES:
Pediatric participants: Brain volume score on MRI at admission and 24 hours (+/- 6 hours) post-randomization, if MRI is available | Measured at baseline and 24 hours post randomization
  Detected by MRI
Pediatric participants: 2. Number of minutes of electrographic seizures within the first 12 hours after DON administration | Measured through 12 hours post infusion
  Detected by continuous EEG monitoring
Pediatric participants: EEG power analysis | Measured at baseline and through 12 hours post infusion
  Detected by 30 minute EEG samples analyzing power at baseline and 3, 6, and 12 hours post infusion
Pediatric participants: EEG amplitude analysis | Measured at baseline and through 12 hours post infusion
  Detected by 30 minute EEG samples analyzing amplitude at baseline and 3, 6, and 12 hours post infusion
Pediatric participants: EEG frequency analysis | Measured at baseline and through 12 hours post infusion
  Detected by 30 minute EEG samples analyzing frequency at baseline and 3, 6, and 12 hours post infusion
Pediatric participants: Transcranial Doppler (TCD) phenotype flow velocities | Measured through 24 hours post infusion
  Detected by TCD at 4H and 24H post infusion
Pediatric participants: Cerebrospinal Fluid Metabolic Profile | Measured through 4 hours post infusion
  Detected by LP at baseline and 4H (+ or - 2H) post DON infusion

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Postels, MD, Principal Investigator — Children's National Research Institute
Locations (2):
- Malawi (2):
  - Ndirande Research Clinic, Blantyre
  - Queen Elizabeth Central Hospital, Blantyre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nampota-Nkomba N, Nyirenda OM, Mallewa J, Chimalizeni Y, Dzabala N, Fay MP, Gopalakrishnan M, Laurens MB, O'Brien NF, Miller LH, Pierce SK, Riggle BA, Postels DG. DON in pediatric cerebral malaria, a phase I/IIA dose-escalation safety study: study protocol for a clinical trial. Trials. 2024 Jan 26;25(1):87. doi: 10.1186/s13063-023-07808-w. PMID 38279124